CLINICAL TRIAL: NCT00448903
Title: Multicentric, Randomized, Double-blind, Controlled Clinical Trial to Assess the Efficacy and Safety of Bemiparin Sodium as Treatment of Diabetic Foot Ulcers
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of Sodium Bemiparin for Treatment of Diabetic Foot Ulcers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rovi Pharmaceuticals Laboratories (Industry)
Responsible Party: Rovi Pharmaceuticals Laboratories, Medical Department
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ROV-BEM-2006-01; 2006-005201-60
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2010-05

CONDITIONS: Foot Ulcer, Diabetic
Keywords: diabetic; foot; ulcer; bemiparin; neuropathy; neuroishemic; diabetes
MeSH Terms: conditions — Diabetic Foot; Ulcer; Diabetes Mellitus | interventions — bemiparin; Ro 11; dexketoprofen trometamol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Bemiparin
  Interventions: Drug: Bemiparin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bemiparin — Bemiparin sodium
  Other Names: RO-11; Hibor; Zibor; Ivor; Badyket; Ivorat; Ivormax; Entervit
  Arms: A
Drug: Placebo — Sodium Chloride 0,9%
  Other Names: Sodium Chloride; physiological saline
  Arms: 2

SUMMARY:
Chronic foot ulcers are a common, severe and expensive complication in patients with diabetes and often causes lower-extremity amputation. The aim of this study is to evaluate the effect of bemiparin as treatment of diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old who have given their informed consent to participate in the study.
* Patients with type I or II Diabetes Mellitus (ADA Criteria).
* Presence of chronic neuropathic inframalleolar diabetic foot ulcer (starting at least 2 months before), grade I or II on Wagner Classification, without significant improvement (reduction of ulcer area > or = 25%) within the past 15 days prior to inclusion.
* Ulcer size equal or bigger than 0.64 cm2 using the following formula: [Major axis] x [Minor axis]
* Ankle-brachial index (ABI) > or = 0,7

Exclusion Criteria:

* Patients with clinical symptoms of limb-threatening or life-threatening infection
* Presence of bone exposure at the bottom of the ulcer and/or bone palpation by catheter and/or presence of radiological signs of pathological fractures and/or bone sequesters
* Ankle-brachial index (ABI) <0,7
* Subjects with arterial calcification (ABI > 1,3) with negative tibial and foot pulse that for any cause the Toe/Arm index (T/A) cannot be measured by plethysmography (photoplethysmography or strain-gauge)
* Subjects with arterial calcification (ABI > 1,3) with negative tibial and foot pulse and with T/A index < 0,55 measured by plethysmography (photoplethysmography or strain-gauge)
* Patients with hematological disorders, organic lesions susceptible to bleeding (e.g. active peptic ulcer, stroke, aneurysms), severe arterial hypertension (systolic blood pressure over 200 mmHg and/or diastolic blood pressure over 120 mmHg).
* Patients with severe renal failure (creatinine clearance <30 ml/min) or hepatic insufficiency (AST and/or ALT values >5 times the normal value established by the reference ranges of the local hospital laboratory).
* Patients with connective tissue disease
* Acute bacterial endocarditis or slow endocarditis.
* Patients with antithrombin deficit and C and S protein deficit.
* Patients with HbA1C > 12%.
* Women who are pregnant or breast-feeding, or with the possibility of becoming pregnant during the study.
* Known hypersensitivity to LMWH, heparin or substances of porcine origin.
* Patients with a history of heparin-induced thrombocytopenia.
* Patients on treatment with anticoagulant therapy at inclusion time or in the past 15 days.
* Patients on treatment with pentoxifiline at inclusion time or in the past 30 days.
* Patients on treatment with systemic corticosteroid or immunosuppressive therapy at inclusion time or in the past 3 months.
* Patients on treatment with beclapermin at inclusion time or in the past 15 days.
* Patients that have suffered a revascularization or endovascular surgery two months prior to inclusion
* Patients with a life expectancy less than 6 months.
* Patients that cannot complete the scheduled follow-up visits or are not able to complete the study period.
* Patients who are participating in another clinical trial or have done it in the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2007-03; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
total healing with intact skin or a significant improvement defined as a reduction of ulcer area > or = 50% or one degree reduction on Wagner Classification. | 90 day

SECONDARY OUTCOMES:
incidence of major bleeding and the incidence of adverse events. | 210 day

CONTACTS AND LOCATIONS:
Overall Officials: JR March, MD, Study Chair — Getafe Hospital, E-28905 Getafe (Madrid) Spain; J Marinel-lo, MD, Study Chair — Mataró Hospital, E-08304 Mataro (Barcelona) Spain; R Gómez Medialdea, MD, Study Chair — Virgen de la Victoria Hospital, E-29010 Malaga, Spain
Locations (6):
- CROATIA, Zagreb, Croatia
- POLAND, Warsaw, Poland
- ROMANIA, Timișoara, Romania
- RUSSIA, Saint Petersburg, Russia
- SERBIA, Belgrade, Serbia
- SPAIN, Madrid, Spain